CLINICAL TRIAL: NCT00582348
Title: Physical Activity and Inactivity in Lung Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 05-094; Grant # CA115212
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer Survivors
Keywords: Lung Cancer; Survivor; Lung
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to learn how often lung cancer survivors exercise. We also want to learn what helps people to be active or prevents them from being active. Learning this will help us to expand services for lung cancer survivors.

DETAILED DESCRIPTION:
Despite the potential benefits of physical activity, particularly for cancer survivors with comorbid pulmonary and cardiac conditions, no previous research has examined the physical activity levels of lung cancer survivors, an underrepresented subpopulation in cancer survivorship research. We address this research gap in the current study, in which a random sample of 200 lung cancer survivors will complete a comprehensive telephone interview or use self-report to complete a questionnaire focusing on physical activity, related covariates, and preferences regarding physical activity counseling and interventions. We estimate the total time for the completion of the interview or self-report questionnaire to be 45-60 minutes. This study will be conducted with survivors of primary lung cancer who are from 1 to 5 years posttreatment and were treated at Memorial Sloan-Kettering Cancer Center (MSKCC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary Stage IA or IB NSCLC;
* Underwent surgical resection for NSCLC at MSKCC;
* From 1 to 5 years post-treatment for NSCLC prior to study recruitment;
* No evidence of disease (NED) at the time of recruitment;
* Can be reached by telephone;
* Able to provide informed consent.

Exclusion Criteria:

* Undergoing active antineoplastic treatment;
* Major psychopathology or cognitive impairment likely in the judgment of the investigator to interfere with participation and compliance with the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible lung cancer survivors will be identified by the Thoracic DMT Data Manager from the Thoracic Surgical Database.
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2005-09; Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
The primary outcomes of this study are physical activity levels and preferences regarding physical activity counseling and interventions | 45-60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center website — http://www.mskcc.org